CLINICAL TRIAL: NCT01758393
Title: A Randomized Trial of Glucocorticoids in Patients With IgG4-Related Disease
Brief Title: Glucocorticoids in Patients With IgG4-RD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-GC-IgG4RD
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: IgG4-related Disease
Keywords: IgG4-related disease; IgG4-RD
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medium Dose (Experimental): Patients are treated with prednisone or equivlent at doseage of 0.5-0.6 mg/kg/d (max 40mg daily) for 3 weeks, then tapering gradually to 15mg/d in 3 months.
  Interventions: Drug: Prednisone
- High Dose (Experimental): Patients are treated with prednisone or equivlent at doseage of 0.8-1.0 mg/kg/d (max 60mg daily) for 3 weeks, then tapering gradually to 15mg/d in 3 months.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone

SUMMARY:
This is a randomized, open-label, single-center clinical trial to compare the efficacy and safety profile for medium-dose versus high dose glucocorticoid in patients with IgG4-related Disease. Patients will be followed for three months to measure the primary outcome and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18-70 years old with informed consent
* Patients with IgG4-RD:

  1. swelling, sclerosing and inflammatory involvement of one or more organ, including sclerosing pancreatitis, sclerosing cholangitis, inflammatory pseudotumors, retroperitoneal or mediastinal fibrosis, interstitial nephritis, hypophysitis, sclerosing dacryoadenitis, sialadenitis, inflammatory aortic aneurysm, lymphadenopathy, or other inflammatory conditions;
  2. elevated serum IgG4 (>1.35 g/L)
  3. histopathologic features of fibrosis and/or lymphocytic and polyclonal plasma cell infiltration (and IgG4+ plasma cells on immunohistology when performed);
  4. exclusion of other diseases.

Exclusion Criteria:

* Previously or currently received glucocorticoid and(or) immunomodulator
* Pregnancy or lactating
* Concurrent severe and/or uncontrolled and/or unstable diseases
* Patient with malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-01 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Complete Response | 3 months
  Complete Response(CR) is defined as resolution of clinical manifestations, biochemical tests (C-reactive Proteins and IgG or IgG4 levels), and imaging studies.

SECONDARY OUTCOMES:
Disease Response | 3 months
  Disease Response is measured by IgG4-RD Responder Index(IgG4-RD RI) and defined as:
  * Improvement of > 2 points in the IgG4-RD RI over baseline
  * No disease flares, as assessed by the IgG4-RD RI.
Adverse Effect | 3 months
  Treatment-related adverse effect, including glucocorticoid-induced diabetes mellitus and infections.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, MD, Principal Investigator — Deptment of Rheumatology, Peking Union Medical College Hospital; Fengchun Zhang, Study Chair — Deptment of Rheumatology, Peking Union Medical College Hospital
Locations (1):
- Deptment of Rheumatology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China